CLINICAL TRIAL: NCT06683092
Title: Restarting Triple Therapy With Robust Monitoring for Adverse Events (RETRIAL)
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Johns Hopkins University (Other); Massachusetts General Hospital (Other); National Jewish Health (Other); Indiana University (Other); Children's Hospital Colorado (Other); University of Kansas Medical Center (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Gregory Sawicki, Co-Chair of Success with Therapies Research Consortium, Boston Children's Hospital
Other Study IDs: IRB-P00050262
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
Keywords: patient care; adverse events; monitoring
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — serum, plasma, white blood cells, stool, sputum, DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RETRIAL-Mental Health: People with CF ages 6 and up with a history of new or worsening mental health symptoms (such as depression, anxiety, mood, sleep) while on elexacaftor/tezacaftor/ivacaftor (ETI) requiring discontinuation or change from standard dosing who start taking vanzacaftor/tezacaftor/deutivacaftor (VTD).
  Interventions: Other: RETRIAL-Mental Health
- RETRIAL-Neuro: People with CF from RETRIAL-Mental Health who experienced new/worsening neurocognitive symptoms (such as brain fog or memory problems) while taking elexacaftor/tezacaftor/ivacaftor (ETI).
  Interventions: Other: RETRIAL-Neuro
- RETRIAL-Liver: People with Cystic Fibrosis ages 6 and up with a history of drug-induced liver injury (such as elevated liver enzymes) attributed to elexacaftor/tezacaftor/ivacaftor (ETI) requiring dose modification or discontinuation who start taking vanzacaftor/tezacaftor/deutivacaftor (VTD).
  Interventions: Other: RETRIAL-Liver

INTERVENTIONS:
Other: RETRIAL-Mental Health — Participants will complete: daily diaries for 6 weeks, from about 2 weeks prior to starting VTD to about 4 weeks after; biweekly surveys, from about 2 weeks prior to starting VTD to 6 months after, and 2 quarterly surveys (at 9mo and 12mo post-initiation of VTD).
  Groups: RETRIAL-Mental Health
Other: RETRIAL-Liver — Participants may have a research liver function test done prior to starting VTD and 28 days after, if not done clinically.
  Participants will complete surveys: before starting VTD, a month after, and quarterly (at about 3, 6, 9, and 12 months) following VTD initiation.
  Groups: RETRIAL-Liver
Other: RETRIAL-Neuro — Participants will complete a neurocognitive assessment prior to starting VTD and 28 days after.
  Groups: RETRIAL-Neuro

SUMMARY:
RETRIAL is a multi-site observational study of people with Cystic Fibrosis (PWCF) ages 6 and up starting the new triple-therapy modulator (vanzacaftor/tezacaftor/deutivacaftor (VTD)), after having experienced neuropsychiatric events and/or liver injury while taking elexacaftor/tezacaftor/ivacaftor (ETI) that resulted in a modification or discontinuation of standard ETI dosing.

DETAILED DESCRIPTION:
RETRIAL is a prospective, longitudinal, observational, multi-site study of people with Cystic Fibrosis (PWCF) ages 6 and up who had to either change how they took or stop taking elexacaftor/tezacaftor/ivacaftor (ETI) due to new or worsening mental health/cognitive symptoms (such as depression, anxiety, mood, sleep, and/or brain fog/memory problems) and/or liver issues (elevated liver enzymes) while taking the standard dose, and who plan to start taking vanzacaftor/tezacaftor/deutivacaftor (VTD).

ELIGIBILITY:
Inclusion Criteria:

RETRIAL-Mental Health:

* PWCF age 6 years and up (if age is < 12 years old, the PWCF's caregiver will complete daily diaries and surveys; see "Caregiver Participant Inclusion Criteria" below)
* Eligible for VTD and intending to take it
* Experienced new or worsening mental health symptoms after initiating ETI, which led to one of the following changes in treatment to currently taking:

  1. No modulators
  2. A modulator other than ETI
  3. A flipped dose of ETI
  4. A reduced dose of ETI
* Willing to delay first VTD dose for short period of time to complete the Baseline assessments
* Has access to a smart device (phone, tablet, etc.) capable of receiving messages with survey links
* Is English-speaking.

RETRIAL-LIVER:

* A person with CF age 6 years and up
* Eligible for VTD and intending to take it
* Experienced drug-induced liver injury (as defined by local care team) after initiating ETI, which led to one of the following changes in treatment to currently taking:

  1. no modulators; or
  2. a modulator other than ETI; or
  3. a reduced or altered dose of ETI;
* Willing to delay first VTD dose for short period of time to complete the Baseline assessments
* Has access to a smart device (phone, tablet, etc.) capable of receiving messages with survey links
* Is English-speaking.

Exclusion Criteria:

RETRIAL-Mental Health:

* Cannot access VTD
* Currently, or prior history of, taking VTD
* Unable or unwilling to follow protocol
* If <12 years old, having another <12-year-old person in the same household consented into the study
* Is actively listed on any transplant list, or within 3 months post-transplant surgery
* Is currently pregnant (test not required)
* Anticipated change in CF Care Centers in the next 6 months
* Any situation that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data.

RETRIAL-LIVER:

* Cannot access VTD
* Currently, or prior history of, taking VTD
* Unable or unwilling to follow protocol
* If <12 years old, having another <12-year-old person in the same household consented into the study
* Any severe, decompensated liver disease (e.g. Child-Pugh, Class C)
* Is actively listed on any transplant list, or within 3 months post-transplant surgery (any organ), or history of liver transplant
* Is currently pregnant (test not required)
* Anticipated change in CF Care Centers in the next 6 months
* Any situation that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data.

Caregiver Participant:

Inclusion Criteria:

* Is a primary, daily caregiver of a person with CF under the age of 12 enrolled in the study
* Has access to smart device (phone, tablet, etc.) capable of receiving messages with survey links
* Is able to read and complete surveys and Daily Diary in English.

Exclusion Criteria:

- Any situation that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female and male people with CF ages 6 and older who are not able to tolerate the standard dose of ETI due to either new/worsening mental health symptoms and/or drug-induced liver injury.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
RETRIAL-Mental Health (1st objective - discontinuation): one-year incidence of discontinuation or change from VTD standard dosing due to new/worsening mental health symptoms. | Baseline to Month 12
  Discontinuation or change from VTD standard dosing due to mental health symptoms at any time during the one-year follow-up as reported in either: daily diaries, biweekly or quarterly surveys, or chart review.
RETRIAL-Mental Health (2nd objective - symptoms): proportion of participants that experience any worsening in mental health symptoms during the 6-month follow-up | Baseline to Month 6
  Change from baseline that exceeds the minimally-important difference (MID) / minimally-important change (MIC) within the first 6 months after starting VTD in any of the following patient-reported outcome measures: (1) depression (PHQ-8 or PROMIS depression parent proxy), (2) anxiety (GAD-7 or PROMIS anxiety parent proxy), (3) anger and irritability (PROMIS-anger or PROMIS-anger parent proxy), (4) cognitive functioning (PROMIS- cognitive function or PROMIS-cognitive function parent proxy), (5) sleep disturbance (PROMIS-sleep disturbance or PROMIS-sleep disturbance parent proxy).
RETRIAL-Mental Health (3rd objective - RETRIAL-Neuro): proportion of participants that have a worsening on the NIH Toolbox's Fluid Cognition Composite score at 1 month follow-up. | Baseline to Day 30
  Decrease in age-adjusted standard score from baseline to 1 month on the NIH Toolbox's Fluid Cognition Composite Score (a performance-based neurocognitive measure) that exceeds MIC ≥ 7.5 points, signifying a worsening in function.
RETRIAL-Liver: one-year incidence of drug-induced liver injury (DILI) with VTD, defined by expert consensus after review of clinical and laboratory data. | Baseline to Month 12
  Positive DILI diagnosis, including those characterized as "likely," "probable," and "highly probable," as reviewed by a hepatology panel of three experts who assign these likelihood scores based upon review of case report forms, including a specific clinical narrative and laboratory values assessing for other potential etiologies.

SECONDARY OUTCOMES:
RETRIAL-Mental Health (1st objective - discontinuation): one-year incidence of discontinuation or change from VTD standard dosing due to any reason. | Baseline to Month 12
  Reported discontinuation or change from VTD standard dosing due to any reason during the one-year follow-up as reported in either: daily diaries, biweekly or quarterly surveys, or chart review.
RETRIAL-Mental Health (2nd objective - symptoms): proportion of participants that experience worsening of _each_ mental health symptom during the 6-month follow-up. | Baseline to Month 6
  Change from baseline that exceeds the MID/MIC of new/worsening symptoms within the first 6 months after starting VTD for _each_ of the following patient-reported outcomes: (1) depression (PHQ-8 or PROMIS depression parent proxy), (2) anxiety (GAD-7 or PROMIS anxiety parent proxy), (3) anger and irritability (PROMIS-anger or PROMIS-anger parent proxy), (4) cognitive functioning (PROMIS- cognitive function or PROMIS-cognitive function parent proxy), (5) sleep disturbance (PROMIS-sleep disturbance or PROMIS-sleep disturbance parent proxy).
RETRIAL-Mental Health (3rd objective - RETRIAL-Neuro): proportion of participants that have a worsening of _each_ of the NIH Toolbox's cognition domain score at 1 month follow-up. | Baseline to Month 1
  Decrease in age-adjusted standard score from baseline to 1-month that exceeds MIC ≥ 7.5 points for _each_ of the following domains: (1) Flanker, (2) Dimensional Change Card Sort (DCCS), (3) Picture Sequence Memory Test (PSMT), (4) List Sorting, (5) Pattern Comparison.
RETRIAL-Liver: one-year incidence of discontinuation or change from VTD standard dosing due to patient-reported or medical team-documented concerns for liver injury. | Baseline to Month 12
  Reported discontinuation or change from VTD standard dosing due to concerns for liver injury during the one-year follow-up as reported in either: 28-day or quarterly surveys, chart review, or case report forms.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Georgiopoulos, MD, Principal Investigator — Massachusetts General Hospital; CJ Bathgate, PhD, Principal Investigator — National Jewish Health; Janis Stoll, MD, Principal Investigator — Washington University at St. Louis
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Nemours Children's, Wilmington, Delaware
  - Nemours Children's, Jacksonville, Florida
  - Nemours Children's, Orlando, Florida
  - Nemours Children's, Pensacola, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Bloomington, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University at St. Louis, St Louis, Missouri
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No